CLINICAL TRIAL: NCT05502705
Title: Effects of Intravenous Lidocaine on Serum BDNF, NGF, miRNA-206 and miRNA-98 in Elderly Patients Undergoing Abdominal Surgery Under General Anesthesia
Brief Title: The Effect of Intravenous Lidocaine on Postoperative Cognitive Function in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Yujingfang202201
Record Dates: First submitted 2022-07-25; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Organ Protection
Keywords: Postoperative cognitive dysfunction; Lidocaine; Brain-derived neurotrophic factor; Nerve growth factor; miRNA-206; miRNA-98
MeSH Terms: conditions — Postoperative Cognitive Complications; Hereditary Sensory and Autonomic Neuropathies | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Experimental): Intravenous bolus of 1.5 mg/kg of lidocaine followed by a continuous infusion of 3.0 mg/kg for the first hour, 1.5 mg/kg for the second hour, 0.7 mg/kg until the end of the surgery.
  Interventions: Drug: Lidocaine
- Normal saline (Placebo Comparator): Normal saline administered as a bolus and an infusion with identical volume and rate changes as the treatment group.
  Interventions: Other: Normal saline (NS)

INTERVENTIONS:
Drug: Lidocaine — Intravenous bolus of 1.5 mg/kg of lidocaine followed by a continuous infusion of 3.0 mg/kg for the frst hour, 1.5 mg/kg for the second hour, 0.7 mg/kg until the end of the surgery
  Arms: Lidocaine
Other: Normal saline (NS) — Patients are received equal volumes of saline intravenously until the end of the surgery
  Arms: Normal saline

SUMMARY:
The purpose of this study is to investigate the efficacy of intravenous lidocaine on BDNF, NGF, miRNA-206 and miRNA-98 in serum in elderly patients undergoing abdominal surgery under general anesthesia.

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction (POCD) is a major complication following surgeries and anesthesia, especially in elderly individuals. Lidocaine, an inexpensive, widely available, and relatively safe compound, is a local anesthetic that readily crosses the blood-brain barrier. Intravenous lidocaine can reduce the incidence of POCD. However, the mechanism is still unclear.

Brain-derived neurotrophic factor (BDNF) and nerve growth factor (NGF), which are regulated by miRNA-206 and miRNA-98 respectively, play a key role in learning, memory, and cognition. Previous studies have shown that the levels of BDNF and NGF can be improved by lidocaine.

The objective of this study is to investigate the efficacy of intravenous lidocaine on the incidence of early POCD, and the levels of BDNF, NGF, miRNA-206 and miRNA-98 in elderly patients undergoing abdominal surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients were scheduled by following abdominal surgery under general anesthesia
* Aged 65 - 80 years
* ASA physical status Ⅱ-Ⅲ

Exclusion Criteria:

* Severe heart, pulmonary, hepatic and renal insufficiency
* History of neurological diseases (including Alzheimer's disease and stroke history)
* Psychological disorder, and drug or alcohol abuse
* History of anesthesia and surgery
* psychiatric illness
* Unwillingness to comply with the protocol or procedures
* Allergic to lidocaine
* Mini-Mental State Examination (MMSE) score<23 before surgery

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline BDNF at 1, 3 days after surgery | at preoperation,1 and 3 days postoperation
  Venous blood samples were sampled before anaesthesia induction and 1, 3 days after surgery for the BDNF by using Enzyme-linked immunosorbent assay.
Changes from Baseline NGF at 1, 3 days after surgery | at preoperation,1 and 3 days postoperation
  Venous blood samples were sampled before anaesthesia induction and 1, 3 days after surgery for the NGF by using Enzyme-linked immunosorbent assay.
Changes from Baseline miRNA-206 at 1, 3 days after surgery | at preoperation,1 and 3 days postoperation
  Venous blood samples were sampled before anaesthesia induction and 1, 3 days after surgery for the miRNA-206 by using PCR.
Changes from Baseline miRNA-98 at 1, 3 days after surgery | at preoperation,1 and 3 days postoperation
  Venous blood samples were sampled before anaesthesia induction and 1, 3 days after surgery for the miRNA-98 by using PCR.

SECONDARY OUTCOMES:
Changes from Baseline mini-mental state examination (MMSE) at 1, 3 days after surgery | at preoperation,1 and 3 days postoperation
  MMSE was performed

OTHER OUTCOMES:
Postoperative cognitive dysfunction (POCD) | at preoperation,1 and 3 days postoperation
  the incidence of POCD

IPD SHARING:
Plan to Share IPD: Undecided